CLINICAL TRIAL: NCT00073099
Title: Digital Image Based Determination of Ocular Surface Vital Dye Staining
Brief Title: Digital Photography to Evaluate Dry Eye
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040048; 04-EI-0048
Record Dates: First submitted 2003-11-14; First posted 2003-11-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-09-06

CONDITIONS: Eye Disease
Keywords: Dry Eye; Lissamine Green; Fluorescein; Conjunctiva; Cornea; Digital Photography; Corneal and Conjunctival Staining
MeSH Terms: conditions — Eye Diseases; Dry Eye Syndromes; Corneal Diseases

SUMMARY:
Surface eye problems (problems of the cornea and conjunctiva), such as dry eye, are often evaluated using ocular surface staining - the application of a colored dye to the surface of the eye. The physician examines the nature, degree, and pattern of staining on the eye's surface to determine the diagnosis, assess disease severity, and document treatment effects. Grading of ocular surface staining is often used in research studies to measure the response to a treatment or treatment side effects. Therefore, it is critical that the grading methodology be reproducible and sufficiently detailed to detect changes in eye health status. Current evaluation techniques using these dyes are somewhat subjective, however, since they require human assessment and judgment. This study will assess the validity and reliability of digital photography and compare it with standard slit lamp evaluation for analyzing ocular surface dye staining to document surface eye damage in patients with dry eye.

Patients 3 years of age and older with dry eye may be eligible for this study. Participants will have the following tests and procedures:

* Visual acuity: (eye chart) test
* Slit lamp evaluation: Examination of the front part of the eye with a special microscope called a slit lamp biomicroscope. Special dyes derived from vegetables are instilled into the eye to stain the surface of the eye where it is dry and damaged. The doctor then determines the extent of staining. The staining will be repeated within one week of the first examination.
* Digital eye photography: Digital photographs of the eye are taken to aid in assessing the extent of dry eye changes. The camera flashes a bright light for each picture. About 5 to 10 pictures are taken for each eye.

DETAILED DESCRIPTION:
Ocular surface vital dye staining is a measure of ocular surface damage and is frequently used as an endpoint in clinical studies. The identification and development of standardized objective outcome measures for the evaluation of therapeutic intervention of ocular surface disease is an area previously identified as critical to the future of well-designed clinical trials in this area. The Report of the NEI / Industry Workshop on Clinical Trials in Dry Eyes identified, the standardization of clinical tests used to diagnose dry eye states and assess treatment effects, as an area of critical interest. The purpose of this protocol is to determine the suitability of slit lamp biomicroscopic digital photography of ocular surface vital dye staining by comparing it to the current standard procedure, clinical assessment. Digital image-based assessment would have many advantages over current procedures and would apply the appropriate rigor to the evaluation of the anterior segment that has been shown to be an extremely effective method for the evaluation of the extent of posterior segment diseases such as diabetic retinopathy and age-related macular degeneration. Such valid, reproducible, reliable photographic documentation of retinal abnormalities and disease progression has been successfully employed as a primary outcome measure in many large clinical trials. In this protocol, we will compare grading of digital images of ocular surface staining to clinical assessment, facilitating the use of ocular surface vital dye staining as a valid outcome measure in clinical trials.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals with ocular surface dysfunction and/or disease are eligible for inclusion in this study.

Individuals being evaluated or treated for ocular surface disease will be enrolled.

EXCLUSION CRITERIA:

Patients who cannot hold their eyes open long enough for the photographs to be taken or who has a known allergy to sodium fluorescein or lissamine green will be excluded.

Children 2 years of age or younger will be excluded since they will not be able to cooperate for slit lamp photography. Dry eye is exceedingly uncommon in this age group.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-11-14; Study Completion 2007-09-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kim J. The use of vital dyes in corneal disease. Curr Opin Ophthalmol. 2000 Aug;11(4):241-7. doi: 10.1097/00055735-200008000-00005. PMID 10977768